CLINICAL TRIAL: NCT00755339
Title: Understanding the Anatomy and Physiology of the Sensory Experience and Its Role in Generating Tics in Tourette Syndrome
Brief Title: Role of the Sensory Experience in Generating Motor Tics in Tourette Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080215; 08-N-0215
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2016-10-25

CONDITIONS: Tic Disorder; Tourette Syndrome
Keywords: Repetitive TMS (rTMS); Magnetoencephalogram; Transcranial Magnetic Stimulation (TMS); Tourette Syndrome; Tic Disorder; Tourete Syndrome
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will investigate the sensation that many people with Tourette syndrome (TS) experience before they have a motor tic. It will also test whether blocking the sensation causes the tic to stop.

People between 18 and 65 years of age with TS who have at least once tic involving an arm may be eligible for this 3-part study. Those enrolled may participate in all parts or in part 1 or part 2. Those who choose to participate in part 3 must first complete part 2. All must stop taking medication for TS and any other medication that may affect the brain for at least 1 week before the study.

Part 1

After numbing the skin or muscles of the arm or leg where a pre-tic sensation is experienced, the response of the nerves will be tested by asking subjects to rate the strength of the sensation after a pinprick and by stimulating the nerves with small electrical shocks. Then, over the course of approximately one hour, subjects will report pre-tic sensations while their motor tics are counted. The onset of each tic will be identified with EMG, a test using electrodes on the skin to indicate the activity of the muscles.

Part 2

Subjects brain waves are recorded using magnetoencephalography (MEG) while they are experiencing tics andpre-tic sensory experiences. MEG is a test that records magnetic field changes produced by brain activity. Subjects sit in a chair under a dome containing magnetic field detectors. They watch a clock and report the time a sensory experience starts. Tics are recorded with EMG. Later, a standard MRI of the brain (scan using a magnetic field and radio waves) is done to see which parts of the brain produced the activity recorded with MEG.

Part 3

Repetitive transcranial magnetic stimulation (rTMS) is used to try to stop the pre-tic sensations. For TMS, the subject sits in a chair. A wire coil is held on the subject s scalp, and a brief electrical current is passed through the coil, creating a magnetic pulse that stimulates a region of the brain. The goal of this stimulation is to reduce the sensory experience that precedes a tic in one region of the body. During stimulation, the subject hears a click and may feel a pulling sensation on the skin under the coil. There may be a twitch in the muscles of the face, arm or leg. This study uses a pattern of repeated pulses delivered in short bursts. Following each train of pulses, the effect of the stimulation on sensation will be tested by asking the subject to rate the strength of a pinprick and of a vibration. In addition, the nerves are stimulated with small shocks to evaluate the effect of the TMS on nerve activity. To determine the effect of TMS on the pre-tic sensation, subjects are asked to watch a clock and report when they are having a sensory experience. The effect on motor tics will be evaluated by using EMG to indicate the tics.

DETAILED DESCRIPTION:
Objectives:

We will investigate whether the sensory experience that precedes motor tics in Tourette syndrome is generated in the peripheral nervous system and whether it may result from altered sensory gating, and whether it is necessary to generate motor tics.

Study Population:

We will study 100 subjects. Thirty-five individuals with a diagnosis of Tourette syndrome who can describe a sensory experience preceding their tics, and 10 who deny a sensory prodrome for a total of 45 subjects. We will also study 55 Healthy volunteers ages 18-65..

Design: A Two-Part Study

Part I: MEG recording

We will determine the extent to which CNS responses to tactile and auditory stimuli habituate. Subjects will be presented with trains of stimuli, repeated 80 times. At the end of each of these blocks, a questionnaire will ascertain the subject s perception of these stimuli. CNS responses to the stimuli will be recorded using MEG and analyzed first for localization, and then for amplitude and frequency characteristics. Healthy volunteers will be included as a control group.

Part II: rTMS inhibition

We will test whether the sensory experience is necessary for generating a motor tic. We will inhibit the sensory experience using repetitive transcranial magnetic stimulation (rTMS) over the cortical region identified by prior and ongoing imaging studies in our group. Low intensity rTMS will be applied as a control. Sensory experiences and motor tics will be recorded before and after rTMS..

Staged Study:

This will be a staged, exploratory study. In phase 1, we will study 20 adult subjects for part II. Data analysis of this phase will determine whether the procedures are well-tolerated and safe enough to allow for the inclusion of adolescent children, ages 14 and older. Phase 2 will involve completion of both parts, with 20 subjects each.

Outcome Measures:<TAB>

For part II, the outcome measures will be 1) inhibition of the sensory experience, and 2) the relationship between inhibition of sensory and motor phenomena. For part I, the outcome measure will be degree of habituation in TS subjects as compared to that in healthy volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Tourette subjects must be 18-65 years of age of any race, gender, or handedness. They must be able to sit for at least 2 hours and remain at the testing site for up to 8 hours. They must be able to follow instructions and participate in reporting sensory experiences. The upper extremity tic to be studied must occur at least once a minute, but no more frequently than once every 5 seconds. Individuals with comorbid attention deficit disorder (ADD or ADHD) or with obsessive-compulsive disorder (OCD) will not be excluded.

Healthy volunteers must be 18-65 years of age, of any race, gender, or handedness.

EXCLUSION CRITERIA:

1. Inability to stop taking all central-acting medications, including those used to treat tics, for at least one week prior to the study
2. Current use of coumadin, heparin, or lovenox
3. Any additional movement disorder, including tremor, myoclonus, or dystonia
4. A diagnosis of major depression or bipolar disorder
5. Frequent or severe headaches
6. Any history of or current experience of hallucinations
7. Any history of a seizure or epilepsy or a family history of epilespy
8. Any prior brain injury, brain tumor or other lesion, stroke, or surgery
9. A diagnosis of increased intracranial pressure
10. A history of significant heart disease
11. Any history of hearing problems, or abnormal results on auditory testing (part I or II)
12. Any of the following: pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, or shrapnel fragments (part I and II only)
13. Any history of work as a welder or metal worker (part I and II)
14. Current pregnancy
15. Tobacco use (cigarette, chewing, or other) in the month prior to the study (part II)
16. Diagnosis of, treatment for, or self-report of alcohol abuse (alcoholism) (part I)
17. Cocaine use in the year prior to involvement in the study (part I)
18. Use of any medication within one month prior to the study with cholinergic or anticholinergic properties, including (but not limited to): nicotine patch, nicorette gum, atrovent, enablex, toriaz, ditropan, vesicare, detrol, sanctura, artane, Aricept, cogentin, akineton, zanaflex, norflex, flexeril, lomotil, mototen, levsin, razadyne, exelon (part I)
19. Peripheral neuropathy or carpal tunnel syndrome (part I)
20. Inability to hold head still for 10 minutes (part I).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-09-15; Study Completion 2016-10-25

PRIMARY OUTCOMES:
Inhibition of the sensory experience frequency and intensity.

SECONDARY OUTCOMES:
The relationship between inhibition of sensory and motor experiences; and detecting and localizing an electromagnetic signal corresponding to the sensory experience.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aoki KR. Review of a proposed mechanism for the antinociceptive action of botulinum toxin type A. Neurotoxicology. 2005 Oct;26(5):785-93. doi: 10.1016/j.neuro.2005.01.017. Epub 2005 Jul 5. PMID 16002144
- [Background] Alary F, Simoes C, Jousmaki V, Forss N, Hari R. Cortical activation associated with passive movements of the human index finger: an MEG study. Neuroimage. 2002 Mar;15(3):691-6. doi: 10.1006/nimg.2001.1010. PMID 11848712
- [Background] Banaschewski T, Woerner W, Rothenberger A. Premonitory sensory phenomena and suppressibility of tics in Tourette syndrome: developmental aspects in children and adolescents. Dev Med Child Neurol. 2003 Oct;45(10):700-3. doi: 10.1017/s0012162203001294. PMID 14515942